CLINICAL TRIAL: NCT02630576
Title: Neurostimulation and Electromyographs Assessment of th TetraGraph in Healthy Volunteers
Brief Title: Neurostimulation and Electromyographs Assessment of th TetraGraph in Healthy (Volunteers
Acronym: NEAT-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Debrecen (Other)
Responsible Party: Principal Investigator, Tamas Vegh, MD, MD, PhD, University of Debrecen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ADBV-ABS-0214-NEAT-2H; 028605-010/2014/OTIG (Registry Identifier: The Office for Health Authorization and Administrative Procedures (EEKH)); DE RKEB/IKEB4170-2014 (Registry Identifier: Regional and Institutional Ethics Committee, university of Debrecen)
Record Dates: First submitted 2015-05-22; First posted 2015-12-15 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Electromyography; Neuromuscular Monitoring
Keywords: electromyography; neuromuscular blockade

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Men - Left Hand (Experimental): 5 healthy male volunteers undergoing 4 types of neuromuscular stimulation protocols on the left hand
  Interventions: Device: Neuromuscular stimulation
- Men - Right Hand (Experimental): 5 healthy male volunteers undergoing 4 types of neuromuscular stimulation protocols on the right hand
  Interventions: Device: Neuromuscular stimulation
- Women - Left Hand (Experimental): 5 healthy female volunteers undergoing 4 types of neuromuscular stimulation protocols on the left hand
  Interventions: Device: Neuromuscular stimulation
- Women - Right Hand (Experimental): 5 healthy female volunteers undergoing 4 types of neuromuscular stimulation protocols on the right hand
  Interventions: Device: Neuromuscular stimulation

INTERVENTIONS:
Device: Neuromuscular stimulation — Single twitch and train-of-four stimulation protocols will be performed at the randomised side with growing current intensity

SUMMARY:
TetraGraph is a newly developed EMG-based (electromyograph), quantitative, battery-powered neuromuscular monitoring system intended for daily clinical use. The primary aim of this clinical investigation is to examine the applicability (ease of use, equipment need, etc.), repeatability (precision or internal consistency) and performance (signal quality, accuracy of outcome, voltage of stimulation output before and during a stimulus) and tolerability of the Tetragraph device in healthy volunteers.

DETAILED DESCRIPTION:
The primary endpoint will be assessment of the ability of the TetraGraph prototype to deliver neuro-stimulation, and assessment of the ability to acquire muscle action potentials and record these evoked responses on the SD-card. The study will be performed on healthy volunteers - 10 male and 10 female. Testing will be done at two separate stimulation/recording sites: ulnar nerve stimulation/abductor digiti minimi (ADM) muscle recording; and ulnar nerve stimulation/adductor pollices (AP) muscle recording. The side of testing (RIGHT vs. LEFT hand) will be determined a priori and randomly by the principal investigator, such that 10 volunteers each will be tested on the RIGHT and 10 on the LEFT hands. At each stimulating/recording site two stimulation protocols (single twitch stimulation and train-of-four stimulation) will be performed with growing current intensity (10-60 mA (milliAmps), in a 10 mA step-up fashion). Volunteers will rate the tolerability of each stimulation protocols on a visual analogue scale. EMG data will be recorded on the SD card and evaluated off-line.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Volunteer is American Society of Anesthesiology (ASA) physical status I-III (Tabl
* Volunteer has provided written informed consent

Exclusion Criteria:

* Presence of an underlying neuromuscular disease
* Use of medications known to interfere with neuromuscular transmission
* Presence of renal or hepatic disease
* Subject has only one upper extremity
* Subject has open sores at the skin sites needed for electrode application

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Primary performance assessment of TetraGraph device | Subjects will be followed for the time of measurements an expected avarage of one hour
  The primary objective of this study is the assessment of the ability of the prototype to deliver neuro-stimulation, and assessment of the ability to acquire muscle action potentials and record these evoked responses on the SD-card.

SECONDARY OUTCOMES:
Secondary performance assessment of TetraGraph Device | Subjects will be followed for the time of measurements an expected avarage of one hour
  The secondary outcome measures is a composite of several performance data:
  1. Confirmation that the prototype can independently stimulate and record repetitive patterns of neuro-stimulation (1 Hz ST and TOF);
  2. Verify that stimulus artifact will not exceed 2.0 mV( millivolt), nor overlap with the evoked EMG response when a stimulus is applied;
  3. Validate the consistency of delivered stimuli, assessed by repeatability of evoked responses.
  4. Verify delivery of neuro-stimulation at varying currents, from the lowest current that produces an evoked response to the current above which the evoked response no longer increases, at increasing current levels separated by steps of 10 mA;
  5. Determine any difference in recording performance using evoked responses (1 Hz ST, TOF) between recordings at two different hand muscles, the abductor digiti minimi and adductor pollices muscles;
  6. Document consistency of stimulation at constant currents independent of patient age, sex, handedness or

OTHER OUTCOMES:
Safety assessment of TetraGraph device | Subjects will be followed for the time of measurements an expected avarage of one hour
  The safety of Tetragraph device will be assesses by checking the stimulating and recording electrode positions for skin reactions and by establishing the discomfort, if any, associated with nerve stimulation in awake, un-medicated human volunteers. Assessment will be made using an 11-point visual analog score (VAS) scale, anchored with 0 (representing no distress) and 10 (representing the worst distress ever experienced) (Table I). These VAS scores will be compared to those reported in the literature.

CONTACTS AND LOCATIONS:
Overall Officials: Bela Fulesdi, MD,PhD,DSci, Principal Investigator — UNIVERSITY OF DEBRECEN FACULTY OF MEDICINE Department of Anesthesiology and Intensive Care Debrecen, Hungary, 4032
Locations (1):
- University of Debrecen, Debrecen, Hungary

REFERENCES:
- [Background] Gatke MR, Viby-Mogensen J, Rosenstock C, Jensen FS, Skovgaard LT. Postoperative muscle paralysis after rocuronium: less residual block when acceleromyography is used. Acta Anaesthesiol Scand. 2002 Feb;46(2):207-13. doi: 10.1034/j.1399-6576.2002.460216.x. PMID 11942873
- [Background] Cammu G, De Witte J, De Veylder J, Byttebier G, Vandeput D, Foubert L, Vandenbroucke G, Deloof T. Postoperative residual paralysis in outpatients versus inpatients. Anesth Analg. 2006 Feb;102(2):426-9. doi: 10.1213/01.ane.0000195543.61123.1f. PMID 16428537
- [Background] Kim KS, Lew SH, Cho HY, Cheong MA. Residual paralysis induced by either vecuronium or rocuronium after reversal with pyridostigmine. Anesth Analg. 2002 Dec;95(6):1656-60, table of contents. doi: 10.1097/00000539-200212000-00033. PMID 12456433
- [Background] Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS. Residual neuromuscular blockade and critical respiratory events in the postanesthesia care unit. Anesth Analg. 2008 Jul;107(1):130-7. doi: 10.1213/ane.0b013e31816d1268. PMID 18635478
- [Background] Murphy GS, Brull SJ. Residual neuromuscular block: lessons unlearned. Part I: definitions, incidence, and adverse physiologic effects of residual neuromuscular block. Anesth Analg. 2010 Jul;111(1):120-8. doi: 10.1213/ANE.0b013e3181da832d. Epub 2010 May 4. PMID 20442260
- [Background] Hemmerling TM, Le N. Brief review: Neuromuscular monitoring: an update for the clinician. Can J Anaesth. 2007 Jan;54(1):58-72. doi: 10.1007/BF03021901. PMID 17197470
- [Background] Brull SJ, Silverman DG. Visual and tactile assessment of neuromuscular fade. Anesth Analg. 1993 Aug;77(2):352-5. doi: 10.1213/00000539-199308000-00024. PMID 8394051
- [Background] Grayling M, Sweeney BP. Recovery from neuromuscular blockade: a survey of practice. Anaesthesia. 2007 Aug;62(8):806-9. doi: 10.1111/j.1365-2044.2007.05101.x. PMID 17635429
- [Background] Claudius C, Viby-Mogensen J. Acceleromyography for use in scientific and clinical practice: a systematic review of the evidence. Anesthesiology. 2008 Jun;108(6):1117-40. doi: 10.1097/ALN.0b013e318173f62f. PMID 18497614
- [Background] Connelly NR, Silverman DG, O'Connor TZ, Brull SJ. Subjective responses to train-of-four and double burst stimulation in awake patients. Anesth Analg. 1990 Jun;70(6):650-3. doi: 10.1213/00000539-199006000-00012. PMID 2160781